CLINICAL TRIAL: NCT04222270
Title: The Impact of Structured Caregiver Peer Support (CaPS) on ART Adherence and Viral Suppression Among Children Living With HIV in Nigeria
Brief Title: Caregiver Peer Support and ART Adherence Among Children
Acronym: CaPS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institute of Human Virology, Nigeria (Other)
Collaborators: University of Maryland, Baltimore (Other); University of Pittsburgh (Other); University of Stellenbosch (Other); University of Georgia (Other)
Responsible Party: Principal Investigator, Tongdiyen Laura Jasper, Continuous Quality Improvement Officer Pediatrics, Institute of Human Virology, Nigeria
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IHVN_IAS_Peds_CaPS
Record Dates: First submitted 2020-01-03; First posted 2020-01-09 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2024-10

CONDITIONS: HIV; Adherence
Keywords: Children; HIV; Caregivers; Peer; Mentors; suppression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Caregiver peer support from Champion caregivers (Peer mentors) to caregivers of unsuppressed children living with HIV (CLHIV) on child care and medication adherence strategies to enhance achievement of viral suppression: Champion Caregivers (Peer Mentors) will be assigned to the intervention arm and will be trained to support 10-15 caregivers for 18 months post enrollment. Champion Caregivers (CCs) be trained using an adapted Mentor-Mother Peer Support curriculum and topics will include pediatric treatment gaps, ARV formulations/dosing, adherence counseling, and virological failure/suppression. Champion caregivers will conduct monthly-to-quarterly 30 min to 1 hr clinic-aligned caregiver group training sessions and home visits at least once quarterly, targeting Child living with HIV (CLHIV) adherence, age-appropriate disclosure, and keeping clinic appointments. The intervention arm will in addition to peer support intervention, receive routine standard of care at the health facility.
  Interventions: Behavioral: Champion Caregiver peer mentoring support to caregivers on child care and medication adherence to enhance achievement of viral suppression
- Control (No Intervention): Unsuppressed Children living with HIV and their caregivers recruited in the control arm will receive no champion caregiver peer support intervention but will continue to receive the standard of care at their health facilities which include routine care, including age-appropriate antiretroviral therapy and clinic appointments (typically every 2-3 months). Routine, albeit brief (5-10 min) adherence counselling is provided to CLHIV/caregivers by trained healthcare workers (HCWs) at every visit. In Nigeria, routine VL is done at 6 months post-ART initiation and repeated 12 months post- initiation 20. VL is done yearly thereafter for suppressed clients. Those unsuppressed receive 3-months' enhanced adherence counselling (EAC) (15-30 min) by Healthcare workers, with intensified appointment schedules and repeat VL upon EAC completion. This rigorous intervention continues until viral suppression is achieved or ART is switched; drug resistance testing (DRT) is not routine.

INTERVENTIONS:
Behavioral: Champion Caregiver peer mentoring support to caregivers on child care and medication adherence to enhance achievement of viral suppression — Caregiver to caregiver peer support intervention through group/one-on-one education and counselling
  Arms: Intervention

SUMMARY:
Adherence for children living with HIV is a by-proxy phenomenon dependent on caregivers (parents, relatives or unrelated guardians) who may or may not be living with HIV. The complexity of paediatric formulations and dosing for ART regimens often poses challenges for caregivers, making ART administration and achievement of viral suppression quite a difficult task for young children. Peer support for caregivers presents a potentially feasible and impactful approach to improve ART adherence and facilitate achievement of viral suppression among children. However, there is a scarcity of robust evidence on the impact of caregiver support as a treatment adherence strategy for children.

The study is a two-arm cluster randomized controlled trial that includes 78 unsuppressed children living with HIV (0-10 years old) and their caregivers at six cluster sites in Nigeria. It will:

* Explore facilitators and barriers to ART adherence among young children to develop a caregiver peer mentor training curriculum and interventional programme.
* Test the impact of caregiver peer support, a locally adapted behavioural intervention, to improve adherence and promote achievement of viral suppression among children.

The intervention will target caregivers of children, measuring outcomes at child level after 12 months of follow up. The intervention arm will receive structured caregiver-to-caregiver peer support while the control arm will receive routine standard of care with no such support. The researchers will compare ART drug-pickup rates and viral suppression for children living with HIV at specific time points for both arms.

DETAILED DESCRIPTION:
Study Purpose and Intervention: The purpose of the study is to evaluate the impact of structured peer support (PS) to caregivers in achieving treatment adherence among children living with HIV in Nigeria. The study adopts a behavioral intervention that engages "expert" caregivers (Champion Caregivers) whose CLHIV wards have achieved viral suppression, to provide structured peer support to other caregivers towards achieving treatment adherence (ART drug-pickup adherence and viral suppression) for their CLHIV. Using a previously-tested structured PS model, Champion Caregivers will receive comprehensive skills-training, including counselling techniques and pediatric ART formulations/administration techniques, and will use standardized logbooks to document client interactions.

Study Aims and Objectives Recent data from Institute of Human Virology Nigeria (IHVN)-supported facilities in the study setting show viral suppression averaging 42.5% among CLHIV <10 years and 61% for those 10-19 years old. Clearly, younger children need prioritization for viral suppression interventions. The structured Mentor Mother PS model was successful in improving viral suppression among HIV-infected women in the same study setting. The PS intervention's structure lies in a focused curriculum, standardized schedules, documentation for client interactions, and performance evaluations. Prior programmatic data indicate that 30-40% of CLHIV have lost at least one biological parent by age 10 years. However, especially for double orphans or indigent/ill single parents, relatives/unrelated guardians (who may or may not be HIV-infected) step in as primary caregivers. Sustained support, education and motivation for caregivers is thus important for optimal CLHIV treatment outcomes. Prescription refill/drug pickup has been a useful, convenient and cost-containing measure of ART adherence in prior studies especially in resource-limited settings. Use of integrase inhibitors is at its infancy in Nigeria. Dolutegravir scale-up started in earnest in 2018; as such, there are no appreciable numbers of children on this drug in early 2019. Approximately 92% of children in the target population are on nevirapine or efavirenz-based regimens. The rest are receiving Lopinavir or atazanavir-based regimens. Drug resistance testing (DRT) is not routine and there is currently no in-country capability to test integrase inhibitor resistance. There is currently no available data from randomized trials evaluating caregiver PS interventions for CLHIV adherence and viral suppression. Given the above context and information, investigators propose a two-arm cluster-randomized Caregiver Peer Support (CaPS) trial at 6 clinics and among 96 CLHIV six months-10 years of age.

Study Design, Methods and Research Participants:

CaPS is a two-arm cluster randomized controlled trial to be conducted at secondary healthcare facilities in two neighboring states: Federal Capital Territory (FCT) and Nasarawa State. Secondary facilities are targeted because majority of children and adolescents living with HIV in Nigeria are managed at secondary health facilities.

Site Eligibility Criteria:

* ≥30 CLHIV aged 6 months to 10 years enrolled in care and on ART
* ≥1 on-site staff providing adherence counselling for CLHIV
* Facility management and staff willing to support study activities In FCT and Nasarawa, there are 15 high-volume secondary facilities receiving President's Emergency Plan for AIDS Relief (PEPFAR)-supported pediatric quality improvement (QI) initiatives which do not include caregiver PS. Six of the 15 sites will be randomly-selected and randomly-assigned 1:1 by computer software to receive intervention (Champion Caregiver) PS or standard-of-care only (no caregiver PS).

Sample Size Minimum sample size is 13 CLHIV per cluster x 6 clusters (3 clusters/arm, 66 CLHIV total). This sample size has 80% power to detect a 22% increase (absolute difference) in ART drug pickup rates (73% to 95%), assuming an intra-cluster correlation of 0.03 and coefficient of variation (k) of 0.21. Effect size of +32% was achieved with structured PS among women living with HIV in the same study setting.

After factoring in ~5% for expected mortality rate among Nigerian CLHIV 36, 5% for study withdrawal and 5% for formal transfer rates, the target sample size per cluster is approximately 13 CLHIV (minimum sample size of 13 + an extra 15%). Total target sample size is thus 96 (16 per cluster x 6 clusters).

Data Analysis Plan The effect of champion caregiver peer support intervention on drug pick-up rate would be assessed by comparing the drug pickup rate at the intervention and control groups. Drug pick-up rates will be categorized into poor, fair and good using <80%, 80%-94% and ≥95% pick-up rates respectively. The pattern of the pick-up rate will be described using frequency and percentage distribution. Effect of CC support on CLHIV viral suppression will be examined using a multivariate logistic regression model with generalized estimating equation to account for clustering. First, univariate models will be performed for association between CC support/intensity and viral suppression. Biologically-plausible variables and those changing crude effect size by ≥ 5% will be sequentially added to the multivariate model. Sensitivity analysis with lower VL threshold of <20 copies/ml is planned. Analysis will be performed with SAS software v 9.4.

Participant Recruitment Investigators will recruit pediatric patients aged between 6 months and 10 years enrolled at pediatric ART clinics within the participating PEPFAR-supported healthcare facilities. Research assistants (RAs) will work with the focal person in the pediatric clinic to identify and recruit eligible patients. RAs will approach the parent/caregiver of the eligible participants to obtain consent for participation in the study. With regard to assent, the Nigerian National Health Research Ethics Committee recommends obtaining assent for children 12 years to under 18 years of age. Given the target age group for CaPS (age 6 months to 10 years), assent would not apply to this study. All children enrolled will be required to only have parental consent.

Privacy and Confidentiality, Risks and Benefits, Ethics

1. Privacy measures include having only healthcare workers first approach caregivers and eligible participants for recruitment. As such, only caregivers and participants who wish to be contacted will be contacted for recruitment. To protect participant's privacy, interviews will take place in a private room.
2. Confidentiality measures include the following: Trained research assistants will meet with participants in a private space at the health facility to administer study questionnaires. Access to study data with private/contact information is restricted to only key study staff. Both hard copy and electronic data will be kept locked or with password protection in secured devices or research file cabinets. Protected health information (PHI) and all study data will be kept confidential following local and international privacy guidelines. Participants will be identified with a study ID and forms will be labelled with the participants' ID instead of their name. Data will be abstracted and stored in an electronic database which will be encrypted. De-identified data will be made available to other members of the team, such as the biostatistician, on a need to know basis. Blood samples will be obtained periodically from all participants for viral load measurement throughout the study. The samples will be collected according to an established protocol in the health facility and labeled with the participant ID.
3. Risks: This study is designed to pose only minimal risk to participants. Physical risk is associated with the blood sample collection needed for viral load assessment. Blood draws carry some risk of causing, pain, bruising and infection. Additional psychological risk may be associated with responding to questions on the psychosocial assessment tools and other qualitative interviews. The questionnaires may make a participant feel uncomfortable, stressed or a sense of invasion of privacy. The main risk to subjects is a potential breach in the protection of the participant's private health information. Participation in the study activities may lead to increased perception of stigma among participants which presents a social risk.

   To reduce physical risk, all blood draws will be performed by a trained healthcare professional during clinic visits. Proper clinical practice (gloves, sharp disposal, etc.) and appropriate medical attention to address any emergency that may arise from the blood draws will be made available.

   Psychological risk will be mitigated by ensuring that research staff are trained to be sensitive to the potential for psychological harm. Participants will be informed that their participation is voluntary and that participants have the right to refuse to answer or withdraw from the study at any point.

   Social risk, including stigma, discrimination and violence, associated with participation in the research activities will be minimized by leveraging on safeguards already in place at the healthcare facilities.
4. Benefits Probable benefits of the research for individual participants The aim of the intervention is to improve viral suppression and long-term clinical outcome for children living with HIV. Enrollment in this program will expose caregivers of CLHIV to knowledge and skill-building activities that may lead to improvement in health outcomes of their child/ward.

Data and Safety Monitoring CaPS will develop a Data Safety Monitoring Plan (DSMP) to oversee and ensure the safety of participants' private health information and the validity and integrity of study data. All study personnel will follow the DSMP guidance for managing data to ensure the research data are collected, verified, and entered in an appropriate manner that reflects completeness, integrity, and is analyzable.

ELIGIBILITY:
Inclusion Criteria:

* CLHIV(Child Living with HIV)-Inclusion Criteria:

  * Age 6 months to 10 years
  * On ART for ≥6 months
* Caregiver-Inclusion Criteria:

  * Adult ≥18 to 65 years old (regardless of gender/HIV status/education)
  * Caring for study-eligible child
  * Primary caregiver: adult living in same household as CLHIV, responsible for providing the child's care at home, administering ART and bringing child to clinic

Exclusion Criteria:

* Child Living with HIV-Exclusion Criteria:

  * Child/ward of Champion Caregiver
  * Will not be receiving care at site for ≥12 months
  * Severe/debilitating AIDS-related or-unrelated illness
  * Study baseline VL result is <1,000 copies/ml
* Caregiver-Exclusion Criteria:

  * Not available to participate for ≥6 months. In the setting, CLHIV often have sequential caregivers; Investigators will account for this potential transitional care in 6-month time-periods. In case of caregiver unavailability/demise, another eligible caregiver will be recruited.

Ages: 6 Months to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 96 (Actual)
Dates: Start 2021-12-01 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2023-11-30 (Actual)

PRIMARY OUTCOMES:
Antiretroviral therapy (ART) drug pickup adherence | 18 months study duration
  Primary outcome of ART adherence: assessed by clinic visit-aligned drug-pickups.
  • % drug-pickup = (actual no. drug-pickups/expected no. drug-pickups) x 100, where expected no. pickups based on appointment schedule applicable to period under consideration. Accounts for CLHIV with varying clinic schedules per viral suppression status. "Grace period" of ± 7 days applied to all expected drug-pickup dates regardless of schedule. Pickups outside grace periods considered invalid. Investigators will determine and compare drug-pickup rates at 6/12/18 months post-enrollment.

SECONDARY OUTCOMES:
Rate of viral suppression | 18 months study duration
  Primary outcome of viral suppression is binary: VL<1,000 copies/ml = suppressed; and VL≥1,000 = unsuppressed/treatment failure. Investigators will determine and compare, at 6, 12 and 18 months, proportions of virally-suppressed CLHIV in each arm.
Prevalence of HIV drug resistance | Baseline
  Drug resistance testing would be conducted for all enrolled CLHIV to assess HIV drug resistance of HIV drug resistance of nucleoside reverse transcriptase inhibitors (NRTIs), non-NRTIs (NNRTIs), protease inhibitors and integrase strand transfer inhibitors among CLHIV.

CONTACTS AND LOCATIONS:
Overall Officials: Tongdiyen Jasper, Principal Investigator — Institute of Human Virology, Nigeria
Locations (1):
- Maitama District Hospital, Abuja, Federal Capital Territory, Nigeria

IPD SHARING:
Plan to Share IPD: No